CLINICAL TRIAL: NCT01734473
Title: Casein Protein and Leucine Supplementation to Induce Anabolism in COPD Patients and Healthy Elderly
Brief Title: Casein Protein and Leucine Supplementation in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, PhD, Texas A&M University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2012-0561
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: COPD
Keywords: COPD; Protein synthesis; Protein breakdown; Muscle wasting; Leucine; Hydrolyzed; Casein protein; Carbohydrates
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Muscular Atrophy | interventions — Carbohydrates; maltodextrin; Leucine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Study day 1 (Experimental): Hydrolyzed casein protein. On each study day participants receive one out of 4 protein meals (interventions). The 4 interventions are given in a randomized order.
  Interventions: Dietary Supplement: Hydrolyzed casein protein
- Study day 2 (Experimental): Hydrolyzed casein protein + carbohydrates. On each study day participants receive one out of 4 protein meals (interventions). The 4 interventions are given in a randomized order.
  Interventions: Dietary Supplement: Hydrolyzed casein protein + carbohydrates
- Study day 3 (Experimental): Hydrolyzed casein protein + leucine. On each study day participants receive one out of 4 protein meals (interventions). The 4 interventions are given in a randomized order.
  Interventions: Dietary Supplement: Hydrolyzed casein protein + leucine
- Study day 4 (Experimental): Hydrolyzed casein protein + carbohydrates + leucine. On each study day participants receive one out of 4 protein meals (interventions). The 4 interventions are given in a randomized order.
  Interventions: Dietary Supplement: Hydrolyzed casein protein + carbohydrates + leucine
- Study Day 5 (Experimental): 4 levels of hydrolyzed casein protein + carbohydrates
  Interventions: Dietary Supplement: 4 levels of hydrolyzed casein protein + carbohydrates

INTERVENTIONS:
Dietary Supplement: Hydrolyzed casein protein — Amount provided is based on the fat-free mass of subject
  Other Names: PeptoPro
  Arms: Study day 1
Dietary Supplement: Hydrolyzed casein protein + carbohydrates — Amount provided is based on the fat-free mass of subject
  Other Names: PeptoPro + maltodextrin
  Arms: Study day 2
Dietary Supplement: Hydrolyzed casein protein + leucine — Amount provided is based on the fat-free mass of subject. Leucine (40% of essential amino acid content)
  Other Names: PeptoPro + leucine
  Arms: Study day 3
Dietary Supplement: Hydrolyzed casein protein + carbohydrates + leucine — Amount provided is based on the fat-free mass of subject. Leucine (40% of essential amino acid content)
  Other Names: PeptoPro + maltodextrin + leucine
  Arms: Study day 4
Dietary Supplement: 4 levels of hydrolyzed casein protein + carbohydrates — Amount provided is based on the fat-free mass of subject. The 4 levels are: 0, 0.02, 0.05, 0.15 g casein protein/kg fat free mass/hr. The ratio between protein and carbohydrates is fixed.
  Other Names: 4 levels of PeptoPro + maltodextrin
  Arms: Study Day 5

SUMMARY:
Weight loss commonly occurs in patients with COPD, negatively influencing their quality of life, treatment response and survival. Loss of muscle protein is generally a central component of this weight loss and independently increases mortality. This study will provide relevant clinical information in regards to the anabolic properties of specific dietary substrates and their co-active anabolic effects. Hypotheses: 1) That supplementation of a hydrolyzed casein-based protein meal with the addition of carbohydrates is more anabolic than a hydrolyzed casein-based protein meal without carbohydrates in COPD patients and healthy older adults; 2) That leucine addition to a hydrolyzed casein-based protein meal only enhances the protein anabolic response in COPD patients and healthy older adults when carbohydrates are not added to the protein meal; 3) That COPD patients have a more efficient protein anabolic response to a hydrolyzed casein-based protein meal than healthy older adults.

A fifth study day was added to measure protein requirements of included individuals to be able to interpret their response to the other interventions on the other study days, and to test the hypothesis that subjects with lower protein requirements respond less to intervention with leucine and/or carbohydrates. For the 5th additional test day we will first approach the 10 COPD and 10 healthy subjects who already completed the first 4 study days (and signed the re-contact form) to come back for this extra test day. We will (pre-)screen these subjects by phone for eligibility and check for changes in their recent medical history (with help of the (pre-)screening questionnaires in CRF). If all inclusion criteria are still met, these subjects will be asked to provide a written re-consent. If necessary, we will recruit new subjects who will complete only one of the four test days (i.e. the test day on which the hydrolyzed casein-based protein meal with carbohydrates is provided) and the additional 5th study day.

DETAILED DESCRIPTION:
The study involves 5 study days. The duration of the first 4 study days is approximately 6.5 hours per day and the duration of the 5th study day is approximately 8 hours. On each of the first 4 study days the effect a casein protein meal with or without leucine and carbohydrates will be examined. On the fifth study day the effect of 4 different levels of casein protein and carbohydrate intake by sip feeding (every 20 minutes) is examined.

Also, subjects will receive a mixture of amino acids (little parts of protein) which are a little bit heavier than normal, called stable isotopes. This is the so-called stable isotope method to investigate protein behavior in the body (protein kinetics). Altogether about 75 ml of blood will be drawn per study day to assess outcome measures.

ELIGIBILITY:
Inclusion criteria COPD subjects:

* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lie in supine or elevated position for 5.5 hours
* Diagnosis of moderate to very severe chronic airflow limitation and compliant to the following criteria: Forced Expiratory Volume(FEV1)/Forced Vital Capacity (FVC) < 0.70 and FEV1 < 70% of reference FEV1
* Clinically stable condition and not suffering from a respiratory tract infection or exacerbation of their disease (defined as a combination of increased cough, sputum purulence, shortness of breath, systemic symptoms such as fever, and a decrease in FEV1 > 10% compared with values when clinically stable in the preceding year) at least 4 weeks prior to the first test day
* Shortness of breath on exertion
* Willingness and ability to comply with the protocol, including:

  * Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Inclusion criteria healthy control subjects:

* Healthy male or female according to the investigator's or appointed staff's judgment
* Ability to walk, sit down and stand up independently
* Age 45 years or older
* Ability to lay in supine or elevated position for 5.5 hours
* No diagnosis of chronic airflow limitation and compliant to the following criteria: FEV1/FVC > 0.70 and FEV1 ≥ 80% of reference FEV1
* Willingness and ability to comply with the protocol, including:

  * Adhering to fasting state from 10 pm ± 2h onwards the day prior to each study visit

Exclusion Criteria all subjects:

* Any condition that may interfere with the definition 'healthy subject' according to the investigator's judgment (for healthy control group only)
* Established diagnosis of malignancy
* Established diagnosis of Insulin Dependent Diabetes Mellitus
* History of untreated metabolic diseases including hepatic or renal disorder
* Presence of acute illness or metabolically unstable chronic illness
* Recent myocardial infarction (less than 1 year)
* Any other condition according to the PI or nurse that was found during the screening visit, that would interfere with the study or safety of the patient
* BMI of < 18.5 or ≥ 35 kg/m2
* Dietary or lifestyle characteristics:

  * Use of protein or amino acid containing nutritional supplements within 5 days of first test day
  * Current alcohol or drug abuse
* Indications related to interaction with study products:

  * Known allergy to milk or milk products
* Use of long-term oral corticosteroids or short course of oral corticosteroids 4 weeks preceding first test day
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
* (Possible) pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-11-28 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2015-05-27 (Actual)

PRIMARY OUTCOMES:
Net whole-body protein synthesis | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Change in net whole-body protein synthesis (whole-body protein synthesis - whole-body protein breakdown)
Net whole-body protein synthesis with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Change in net whole-body protein synthesis (whole-body protein synthesis - whole-body protein breakdown) with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)

SECONDARY OUTCOMES:
Whole-body protein synthesis | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Change in whole-body protein synthesis
Whole-body protein breakdown | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Change in whole-body protein breakdown
Splanchnic extraction | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  The amount of amino acids in the protein meal extracted by the splanchnic tissues after intake
Body composition | 1 day
  Difference in muscle mass, fat mass and bone density between COPD patients and healthy older adults
Skeletal and respiratory muscle strength | 1 day
  Difference in handgrip strength and fatigue and maximum inspiratory and expiratory pressure between COPD patients and healthy older adults
Inflammatory mediators | 90 min before protein meal
  C-reactive protein, interleukines
Hormones | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Area under the plasma concentration versus time curve (AUC) of insulin
Glucose | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Peak plasma concentration (Cmax) of glucose
Amino acid concentrations | 0, 15, 30, 45, 60, 90, 120, 150, 180, 210, 240 min post-protein meal
  Peak plasma concentration (Cmax) of amino acids
Whole-body protein synthesis with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Change in whole-body protein synthesis with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)
Whole-body protein breakdown with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Change in whole-body protein breakdown with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)
Splanchnic extraction with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  The amount of amino acids in the protein meal extracted by the splanchnic tissues after intake of 4 different levels of protein (duration of each level: 2 hours) as sip feeding (every 20 minutes)
Hormones with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Area under the plasma concentration versus time curve (AUC) of insulin with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)
Glucose with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Peak plasma concentration (Cmax) of glucose with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)
Amino acid concentrations with different levels of protein intake (Fifth Study Day) | before each sip feeding in the second hour of a level of protein intake ( at 120, 140 and 160 min)
  Peak plasma concentration (Cmax) of amino acids with 4 different levels of protein intake (duration of each level: 2 hours) as sip feeding (every 20 minutes)

OTHER OUTCOMES:
Occurrence of (serious) adverse events | Up to 1 year
  Number of (serious) adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marielle PK Engelen, PhD, Principal Investigator — Texas A&M University
Locations (1):
- Texas A&M University, College Station, Texas, United States

REFERENCES:
- [Derived] Jonker R, Deutz NEP, Schols AMWJ, Veley EA, Harrykissoon R, Zachria AJ, Engelen MPKJ. Whole body protein anabolism in COPD patients and healthy older adults is not enhanced by adding either carbohydrates or leucine to a serving of protein. Clin Nutr. 2019 Aug;38(4):1684-1691. doi: 10.1016/j.clnu.2018.08.006. Epub 2018 Aug 16. PMID 30150004
- [Derived] Jonker R, Deutz NEP, Ligthart-Melis GC, Zachria AJ, Veley EA, Harrykissoon R, Engelen MPKJ. Preserved anabolic threshold and capacity as estimated by a novel stable tracer approach suggests no anabolic resistance or increased requirements in weight stable COPD patients. Clin Nutr. 2019 Aug;38(4):1833-1843. doi: 10.1016/j.clnu.2018.07.018. Epub 2018 Jul 31. PMID 30100106
- See also: PeptoPro — https://www.dsm.com/markets/foodandbeverages/en_US/products/nutraceuticals/peptopro.html